CLINICAL TRIAL: NCT03918577
Title: Caloric Vestibular Stimulation for Modulation of Insight in Obsessive-Compulsive Spectrum Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter J van Roessel, MD PhD, Clinical Assistant Professor, Dept. Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 45068
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder; Body Dysmorphic Disorders; Illness Anxiety Disorder
Keywords: Caloric Vestibular Stimulation; Insight
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Body Dysmorphic Disorders

STUDY DESIGN:
Intervention Model Description: randomized, controlled crossover study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right cold caloric vestibular stimulation (Experimental): OCRD participants in this arm will receive an approx 60 second infusion of distilled cold(4)c water in their right external ear canal, with before and after measures of OCRD symptom severity and insight.
  Interventions: Other: Caloric Vestibular Stimulation
- left cold caloric vestibular stimulation (Experimental): OCRD participants in this arm will receive an approx 60 second infusion of distilled cold(4)c water in their left external ear canal, with before and after measures of OCRD symptom severity and insight.
  Interventions: Other: Caloric Vestibular Stimulation

INTERVENTIONS:
Other: Caloric Vestibular Stimulation — Cold water creates a convection current in the semicircular canal of the vestibular apparatus, leading to brief (<3 min) and typically well tolerated sense of rotational movement. Similar stimulation is routinely used in standard vestibular diagnostic testing.

SUMMARY:
This study investigates whether caloric vestibular stimulation can modulate a measure of insight in obsessive-compulsive spectrum disorders.

DETAILED DESCRIPTION:
Obsessive-compulsive and related disorders (OCRD), including obsessive compulsive disorder and body dysmorphic disorder, are chronic and disabling conditions characterized by recurrent intrusive thoughts and associated compulsive behaviors that affect millions of individuals in the US each year. Individuals affected by OCRD differ in insight, or the degree to which they understand their intrusive thoughts to reflect illness. Impairments in insight limit individuals' motivation to engage in care and predict worse outcome in those who access treatment.

This study seeks to explore whether unilateral stimulation of the vestibular system, which activates cortical areas hypothesized to underlie clinical insight, may beneficially modulate insight in individuals with OCRD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Primary diagnosis of Obsessive-Compulsive Disorder, Body Dysmorphic Disorder, Illness Anxiety Disorder or Somatic Symptom Disorder (excluding "with predominant pain")
* Strongly held OCRD-related concerns meeting BABS score criterion.
* No recent change in psychopharmacological treatment, if any
* Capacity to provide informed consent

Exclusion Criteria:

* Psychiatric or medical conditions (eg, vertigo, history of otological surgery) that might make participation unsafe
* Pregnant or nursing women
* Active or recent substance use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
change in clinical insight as measured by the Brown Assessment of Beliefs (BABS). | 1 hour
  Changes in clinical insight will be rated using the BABS, a gold-standard measure for assessing multiple dimensions of clinical insight across psychiatric disorders. The BABS is a 24 point scale for which scores ≥13 suggest poor or absent insight.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J van Roessel, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- See also: Stanford Medicine Faculty Page — https://med.stanford.edu/profiles/peter-van-roessel
- See also: Rodriguez Lab Website — http://med.stanford.edu/rodriguezlab/research.html